CLINICAL TRIAL: NCT00579540
Title: CCRC: Prevention of Post-Prandial Hypoglycemia Using n-3/n-6 PUFA in PCOS
Brief Title: Compare Effects of Flax Seed Oil, and Fish Oil on Blood Sugar Levels
Acronym: PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200715060
Record Dates: First submitted 2007-12-17; First posted 2007-12-24 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Polycystic Ovarian Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Linseed Oil; Fish Oils; Soybean Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Subject will follow their usual diet for 4 weeks, at week 6 they will be randomized to receive either flax seed oil, fish oil, or soybean oil capsules for 6 weeks.
  Interventions: Dietary Supplement: Flax Seed Oil; Dietary Supplement: Fish Oil; Dietary Supplement: Soybean Oil
- 2 (Active Comparator): Subject will follow their usual diet for 4 weeks, at week 6 they will be randomized to receive either flax seed oil, fish oil, or soybean oil capsules for 6 weeks.
  Interventions: Dietary Supplement: Flax Seed Oil; Dietary Supplement: Fish Oil; Dietary Supplement: Soybean Oil
- 3 (Active Comparator): Subject will follow their usual diet for 4 weeks, at week 6 they will be randomized to receive either flax seed oil, fish oil, or soybean oil capsules for 6 weeks.
  Interventions: Dietary Supplement: Flax Seed Oil; Dietary Supplement: Fish Oil; Dietary Supplement: Soybean Oil

INTERVENTIONS:
Dietary Supplement: Flax Seed Oil — Subject will follow their usual diet for 4 weeks, at week 6 they will be randomized to receive either flax seed oil, fish oil, or soybean oil capsules for 6 weeks. They will take six capsules orally six times a day for a total of six weeks.
Dietary Supplement: Fish Oil — Subject will follow their usual diet for 4 weeks, at week 6 they will be randomized to receive either flax seed, fish oil, or soybean oil capsules for 6 weeks. They will take six capsules orally six times a day for a total of six weeks.
Dietary Supplement: Soybean Oil — Subject will follow their usual diet for 4 weeks, at week 6 they will be randomized to receive either flax seed, fish oil, or soybean oil capsules for 6 weeks. They will take six capsules orally six times a day for a total of six weeks.

SUMMARY:
Flax seed oil, fish oil, and soy bean oil, are commonly recommended supplements for Polycystic Ovarian Syndrome (PCOS). These oils have different chemical structures and biological actions. It is not yet known which of these oils has the most beneficial effects in PCOS patients because they have never been compared to each other head to head. In this study the researchers hope to learn more about the effects of these oils on blood sugar and insulin levels.

DETAILED DESCRIPTION:
The aim is to investigate whether n-3 PUFA's can be used to prevent postprandial hypoglycemia and its unfavorable consequences, such as stimulation of cortisol and adrenal androgen secretion, in women with polycystic ovarian syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Females ages 18-45
* Women who are overweight, and have irregular periods or have been diagnosed with Polycystic Ovarian Syndrome

Exclusion Criteria:

* Use of oral contraceptives
* Impaired glucose tolerance
* Diabetes mellitus, and any other systemic illnesses such as renal, hepatic, gastrointestinal, severe hyperlipidemia and hypertension that require medication
* Schizophrenia
* Having a pacemaker
* Current viral infection
* Smoking alcohol intake (more than 2 drinks/week)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2007-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
We hope to learn more about the effects of fish oil, flax seed oil, and soybean oil, on blood sugar and insulin levels in PCOS patients | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Sidika Kasim-Karakas, MD, Principal Investigator — UC Davis
Locations (1):
- UC Davis, Sacramento, California, United States